CLINICAL TRIAL: NCT01434069
Title: Phase I Trial of Combination of FOLFIRI and SOM 230 in Advanced Gastrointestinal Malignancies
Brief Title: Phase I Trial of Combination of FOLFIRI and SOM 230
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16569; SOM230CUS17T (Other: Novartis)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Gastrointestinal Tumor
Keywords: colon; rectum; small bowel; pancreas; gastric; esophageal; metastatic; unresectable; GI; combination therapy; dose escalation; solid tumor
MeSH Terms: conditions — Digestive System Neoplasms; Neoplasm Metastasis | interventions — Fluorouracil; Leucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Therapy: FOLFIRI and SOM 230 (Experimental): Treatment will be administered on an outpatient basis. FOLFIRI is administered by IV infusion every 2 weeks. The dose should be based on the patient's actual baseline body weight; the dose will be recalculated if there is a weight change of > 10% from baseline.
  SOM 230 will be administered as an intramuscular dose determined by the dosing schema, every 28 days.
  Interventions: Drug: SOM230C LAR; Drug: FOLFIRI Infusion

INTERVENTIONS:
Drug: SOM230C LAR — Participants will be given one LAR dose injected into the muscle of the buttocks by a study nurse about once every 28 days until unacceptable toxicity or progression of the disease.
  Other Names: Pasireotide LAR
Drug: FOLFIRI Infusion — Standard therapy of FOLFIRI
  Other Names: 5-Fluorouracil (5FU), leucovorin (LV), and irrinotecan

SUMMARY:
This is a single-arm, open-label, phase I study of combination therapy with SOM 230 and FOLFIRI. We will utilize a sequential dose-escalation design to define the maximum tolerated dose (MTD) of SOM 230 when combined with standard doses of FOLFIRI.

DETAILED DESCRIPTION:
The goal of this clinical research study is to learn if the study drug SOM 230, also known as Pasireotide long-acting release (LAR), in addition to standard therapy of FOLFIRI (5FU, leucovorin, and irrinotecan) can shrink or slow the growth of gastrointestinal malignancies. The safety of this drug in combination with standard chemotherapy (FOLFIRI) will also be studied. The participant's physical state, changes in the size of the tumor, and laboratory findings taken while on-study will help us decide if Pasireotide LAR is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic/unresectable gastrointestinal malignancies (colon, small bowel, pancreas, gastric and esophageal cancer, etc.) not amenable to curative surgical therapy, for whom FOLFIRI can be considered a standard treatment
* Have had at least 1 prior treatment for all GI tumors except for small bowel adenocarcinoma as FOLFIRI can be considered standard first line therapy for that particular tumor.
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* ≥ 4 weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, Platelets ≥ 100 x 10^9/L, hemoglobin (Hgb) > 9 g/dL
* Adequate liver function as shown by: serum bilirubin ≤ 2 x upper limit of normal (ULN), and serum transaminases activity ≤ 3 x ULN
* Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. Note: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information

Exclusion Criteria:

* Prior treatment with irinotecan. Irinotecan with radiation will be allowed if > 4 weeks.
* Any cytotoxic chemotherapy, radiation, immunotherapy, or any investigational drug within the preceding 3 weeks of starting the study treatment
* History of liver disease, such as cirrhosis or chronic active hepatitis B and C
* History of, or current alcohol misuse/abuse within the past 12 months
* Known gallbladder or bile duct disease, ( ie infection or cholecystitis) acute or chronic pancreatitis
* Have undergone major surgery within 4 weeks prior to study enrollment
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Patients who have been treated at least 4 weeks prior to enrollment, and have a computed tomography (CT) scan or magnetic resonance imaging (MRI) of brain within 4 weeks of enrollment, which shows no evidence of progression of disease in brain, are allowed to enroll.
* Patients with uncontrolled diabetes mellitus defined as hemoglobin A1c (HbA1c) >8% despite therapy or a fasting plasma glucose > 1.5 ULN. Note: At the principal investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
* Symptomatic cholelithiasis
* Have congestive heart failure: New York Heart Association (NYHA) Class III or IV and unstable angina
* History of syncope or family history of idiopathic sudden death
* Sustained or clinically significant cardiac arrhythmias including sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block (Mobitz II or higher atrioventricular nodal block AV)) , patients with prolonged corrected QT interval (QTc) (longer than 470 milliseconds) or a history of acute myocardial infarction within the 6 months preceding enrollment. (The "QT interval" is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle. The "QTc" is the QT interval corrected for heart rate.)
* Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Patients found to have sustained ventricular tachycardia, ventricular fibrillation, advanced heart block (Mobitz II or higher AV nodal block) , prolonged QTc (average longer than 470 milliseconds) in the holter monitor at the screening time. (this only applies to patients in cohorts of 60 mg of SOM 230 or higher)
* Concomitant medication(s) known to prolong the QT interval (patient must be off the drug for 2 weeks to be eligible)
* Presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as: Severely impaired lung function; Any active (acute or chronic) or uncontrolled infection/ disorders; Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
* Known or suspected allergy or hypersensitivity to any component of FOLFIRI, somatostatin analogues or any component of the pasireotide or octreotide long acting release (LAR) formulations
* No active malignancy except for nonmelanoma skin cancer or in situ cervical cancer or treated cancer from which the patient has been continuously disease free more than 5 years
* Women pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control. WOCBP must have a negative serum pregnancy test within 14 days prior to administration of pasireotide. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study
* Unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Average of 6 Months Per Participant
  To determine the maximum tolerated dose (using a standard 3+3 design), of SOM 230 and FOLFIRI.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Average of 6 Months Per Participant
  Evaluate the frequency of toxicities by type and severity, and dose of study drug according to the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.
Number of Participants With Tumor Response | Average of 6 Months Per Participant
  Evaluate the frequency of tumor response by dose cohort according to the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Kim, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States